CLINICAL TRIAL: NCT03125837
Title: Study on the Method of Difficult Airway Prediction Based on Artificial Intelligence
Brief Title: Establishment of Airway Database for Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-076
Record Dates: First submitted 2017-03-13; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Difficult Airway; Artificial Intelligence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Digital photographs of the face and neck
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- general anesthesia: Digital photographs of the face of each patient undergoing general anesthesia with endotracheal intubation

SUMMARY:
Difficult airway is a major reason of anesthesia related injuries with latent life threatening complications. Foresee difficult airway in the preoperative period is vital for the patient's safety. The aim of this study is to develop a computer algorithm that can detect whether the patient is a difficult airway based on photographs form six aspects. This method will be decreased potential complication related to difficult airway and increased patient safety.

DETAILED DESCRIPTION:
Introduction:

The primary purpose of the study is to develop a computer algorithm that can detect whether the patient is a difficult airway based on photographs from six different aspects.

Methods:

This study is divided into two parts. In the first part, we collected the patients' airway assessment score who underwent general anesthesia with endotracheal intubation assessed by an experienced attending anesthesiologists before and after intubation. Evaluation of airway score after tracheal intubation as the gold standard for airway assessment. Digital photographs of the face of each patient in frontal neutral view and in profile neutrals were obtained. Details of the photographs, each corresponding to a facial motion: (1) Frontal, neutral. (2) Frontal, mouth open. (3)Frontal, extreme mouth open and tongue out. (4)Frontal, extreme upper lip bite (5)Profile, neutral. (6) Profile, neutral, maximum head back. The patient's photographs and the airway evaluation score after intubation were input to the computer to train the computer. In the second part, the trained computer was used to evaluate the airway score of the new patient compared with that of the patient after intubation, and calculated the sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* General anesthesia-induced tracheal intubation in patients who undergoing elective surgical patients

Exclusion Criteria:

* Patients with multiple facial injuries Patients who had undergone head or neck surgery Patients who need emergency operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients who underwent general anesthesia with endotracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
the sensitivity of artificial Intelligence to predict difficulty of facemask ventilation and endotracheal intubation | 5 years
  The outcome will be a computer algorithm that can detect whether the patient is a difficult airway based on photographs from six different aspects.Details of the photographs, each corresponding to a facial motion: (1) Frontal, neutral. (2) Frontal, mouth open. (3)Frontal, extreme mouth open and tongue out. (4)Frontal, extreme upper lip bite (5)Profile, neutral. (6) Profile, neutral, maximum head back.

IPD SHARING:
Plan to Share IPD: No